CLINICAL TRIAL: NCT03915899
Title: A Community-Randomized Trial to Reduce HIV Acquisition and Viral Load Among Migrants in Rakai, Uganda
Brief Title: The Welcome Incoming Neighbor (WIN) Community Trial
Acronym: WIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: WIRB20031318
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: HIV

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WIN Intervention (Experimental): WIN Intervention
  Interventions: Behavioral: WIN (Welcome Incoming Neighbor)
- Standard of Care (No Intervention): No WIN intervention.

INTERVENTIONS:
Behavioral: WIN (Welcome Incoming Neighbor) — WINs will conduct active community surveillance to rapidly identify and welcome in-migrants, provide them with information about the availability of CHP, utilize a motivational interviewing approach to encourage CHP adoption, refer in-migrants to free services, and follow-up in-migrants to assess and further encourage engagement in CHP.
  Arms: WIN Intervention

SUMMARY:
Migration is common in rural Africa: in-migrants have higher HIV incidence and prevalence than community residents, but underutilize combined HIV prevention and care services, including voluntary medical male circumcision and antiretroviral therapy, increasing the risks of HIV acquisition and onward transmission. Uptake of combined HIV prevention (CHP) is critical in this vulnerable population. The investigators will conduct a community randomized trial to rapidly identify and link migrants to CHP in rural Uganda; if effective, the intervention could be widely implemented as an important strategy towards HIV epidemic control.

DETAILED DESCRIPTION:
The Rakai Health Sciences Program (RHSP), Uganda, proposes an implementation science community- randomized controlled trial (CRCT) of a novel intervention to newly in-migrated individuals ("Welcome Incoming Neighbor" [WIN]), to optimize in-migrated individuals' rapid linkage to combination HIV prevention (CHP) services. RHSP data show that within the first 36 months after in-migration, compared to residents, HIV-negative in-migrants are at increased risk of HIV acquisition and HIV+ in-migrants underutilize antiretroviral therapy (ART) increasing the risk of onward transmission. The theory-based WIN intervention includes community sensitization and community-based WIN scouts (WINs). WINs will conduct active community surveillance to rapidly identify and welcome in-migrants, provide the in-migrants with information about the availability of CHP and high rates of use by residents (to "normalize" uptake), utilize a motivational interviewing approach to encourage CHP adoption, refer in-migrants to free services, and follow-up in-migrants to assess and further encourage engagement in CHP. Specific Aims: Aim 1: To randomize 40 individually matched communities in a 1:1 ratio to the WIN intervention or control arm. In-migrants aged 15-49 in each arm will undergo a baseline and 2 follow-up surveys at ~18-month intervals. Study end points are CHP coverage rates, HIV incidence in initially HIV-negative in-migrants (n ~3,800 py per arm), and viral load suppression in HIV+ (n ~740 per arm). Aim 2a: To use a mixed methods approach (in-depth interviews, process & survey data) and Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) to (i) guide interim intervention adaptation as necessary; (ii) interpret trial results; and, (iii) translate the research into future action. Aim 2b: To conduct cost studies to provide information on affordability and sustainability. Innovation and Impact: This novel intervention will rapidly engage a vulnerable priority population of in-migrants, to optimize CHP and HIV impact in rural Uganda.

ELIGIBILITY:
Inclusion Criteria:

* Residing in study community

Exclusion Criteria:

* Unable or unwilling to provide informed consent.

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9080 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Antiretroviral Therapy (ART) Coverage as assessed by Proportion of HIV positive Reporting ART Use | 3 years
Male Circumcision Coverage assessed by Proportion of Men Reporting Circumcision | 3 years
Proportion of participants with HIV Viral Suppression | 3 years
Incidence of HIV infection | 3 years
  Rate of New HIV Infections

CONTACTS AND LOCATIONS:
Overall Officials: Maria Wawer, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Rakai Health Sciences Program, Kalisizo, Uganda

IPD SHARING:
Plan to Share IPD: Yes
The Rakai Health Sciences Program (RHSP) has a written policy on the sharing of data and of laboratory specimens. Institutions, groups or researchers who propose to use Rakai data or specimens are required to submit a brief proposal/data request form describing the goals and methods of the proposed analyses. Based on this document and additional discussions with the party(ies) proposing the collaboration, the decision as to whether and/or how to proceed is made by consensus between senior Ugandan and US-based Investigators. The decision takes into account Uganda Ministry of Health directives regarding the maximization of research findings and safeguards regarding misuse, misappropriation or misinterpretation of data. Feasibility, availability of resources (such as Rakai Program analysts' time to help prepare and anonymize data sets to ensure no potential loss of confidentiality), and research importance/priority are also taken into consideration.
Supporting Information: Study Protocol
Time Frame: After Publication of Final Study Outcomes
Access Criteria: Email PI. See plan description.